CLINICAL TRIAL: NCT00721708
Title: Pharmacokinetics of Carnosine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Kyung-Jin Yeum, Scientist, Tufts University
Model: Crossover | Masking: None
Other Study IDs: TMC/TUHS IRB 7737
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Oxidative Stress
Keywords: histidine dipeptides; carnosine; anserine
MeSH Terms: interventions — Red Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Carnosine(450 mg)
  Interventions: Dietary Supplement: pure carnosine
- 2 (Experimental): Beef (150g)
  Interventions: Other: Beef
- 3 (Experimental): chicken (150g)
  Interventions: Other: Chicken
- 4 (Experimental): Chicken broth (obtained from 150 g of chicken breast)
  Interventions: Other: Chicken broth

INTERVENTIONS:
Dietary Supplement: pure carnosine — one time dose of pure carnosine (450 mg)
  Arms: 1
Other: Beef — one time dose, 150 g of beef
  Arms: 2
Other: Chicken — One time dose, 150g of chicken breast
  Arms: 3
Other: Chicken broth — one time dose of chicken broth obtained from 150g of chicken breast
  Arms: 4

SUMMARY:
The absorption kinetics of dietary carnosine (β-alanyl-L-histidine) will be determined in the healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* normal hematological parameters, normal serum albumin, normal liver function, normal kidney function

Exclusion Criteria:

* History of smoking or alcoholism

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Plasma histidine-dipeptide | 0, 30, 60, 100, 180, 240, & 300 min

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Jin Yeum, Ph.D., Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA-Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Result] Yeum KJ, Orioli M, Regazzoni L, Carini M, Rasmussen H, Russell RM, Aldini G. Profiling histidine dipeptides in plasma and urine after ingesting beef, chicken or chicken broth in humans. Amino Acids. 2010 Mar;38(3):847-58. doi: 10.1007/s00726-009-0291-2. Epub 2009 Apr 19. PMID 19381778